CLINICAL TRIAL: NCT00683397
Title: Frankfurt Thrombophilia Registry - Evaluation of Patients With Venous Thromboembolism
Brief Title: Frankfurt Thrombophilia Registry
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. E. Lindhoff-Last, M.D., Cardioangiologisches Centrum Bethanien
Other Study IDs: MAISTHRO Study 93/08
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Venous Thromboembolism
Keywords: assess; prevalence; thrombophilia; common; VTE; risk factors; patients
MeSH Terms: conditions — Venous Thromboembolism; Thrombophilia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum

GROUPS / COHORTS (1):
- A: Patients with acute or previous venous thromboembolism >18 years of age
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Screening of thrombophilia

SUMMARY:
Consecutive patients with acute or previous venous thromboembolism are enrolled in this registry. Using a standardized questionnaire, clinical data detailing venous thromboembolism and contributing VTE risk factors are recorded. Results of technical and laboratory investigations including screening for thrombophilic disorders were additionally entered into the database.

ELIGIBILITY:
Inclusion Criteria:

* Acute or previous VTE

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients with acute or previous VTE >18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2008-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Professor, Principal Investigator — Cardioangiologisches Zentrum Bethanien
Locations (1):
- Cardioangiologisches Centrum Bethanien, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Result] Kraft C, Schuettfort G, Weil Y, Tirneci V, Kasper A, Haberichter B, Schwonberg J, Schindewolf M, Lindhoff-Last E, Linnemann B. Thrombosis of the inferior vena cava and malignant disease. Thromb Res. 2014 Sep;134(3):668-73. doi: 10.1016/j.thromres.2014.07.012. Epub 2014 Jul 18. PMID 25081831
- [Result] Linnemann B, Kraft C, Roskos M, Zgouras D, Lindhoff-Last E. Inferior vena cava thrombosis and its relationship with the JAK2V617F mutation and chronic myeloproliferative disease. Thromb Res. 2012 Jun;129(6):720-4. doi: 10.1016/j.thromres.2011.09.011. Epub 2011 Oct 7. PMID 21982959
- [Result] Schimanski S, Linnemann B, Luxembourg B, Seifried E, Jilg W, Lindhoff-Last E, Schambeck CM. Cytomegalovirus infection is associated with venous thromboembolism of immunocompetent adults--a case-control study. Ann Hematol. 2012 Apr;91(4):597-604. doi: 10.1007/s00277-011-1334-9. Epub 2011 Sep 9. PMID 21913128
- [Result] Luxembourg B, Schmitt J, Humpich M, Glowatzki M, Dressler D, Seifried E, Lindhoff-Last E. Cardiovascular risk factors in idiopathic compared to risk-associated venous thromboembolism: A focus on fibrinogen, factor VIII, and high-sensitivity C-reactive protein (hs-CRP). Thromb Haemost. 2009 Oct;102(4):668-75. doi: 10.1160/TH-09-02-0104. PMID 19806251
- [Result] Luxembourg B, Schmitt J, Humpich M, Glowatzki M, Seifried E, Lindhoff-Last E. Intrinsic clotting factors in dependency of age, sex, body mass index, and oral contraceptives: definition and risk of elevated clotting factor levels. Blood Coagul Fibrinolysis. 2009 Oct;20(7):524-34. doi: 10.1097/MBC.0b013e32832d9b58. PMID 19620844
- [Result] Weingarz L, Schindewolf M, Schwonberg J, Hecking C, Wolf Z, Erbe M, Lindhoff-Last E, Linnemann B. Thrombophilia and risk of VTE recurrence according to the age at the time of first VTE manifestation. Vasa. 2015 Jul;44(4):313-23. doi: 10.1024/0301-1526/a000447. PMID 26314364
- [Result] Linnemann B, Weingarz L, Schindewolf M, Schwonberg J, Weber A, Herrmann E, Lindhoff-Last E. Prevalence of established risk factors for venous thromboembolism according to age. J Vasc Surg Venous Lymphat Disord. 2014 Apr;2(2):131-9. doi: 10.1016/j.jvsv.2013.09.006. Epub 2014 Jan 16. PMID 26993177
- [Result] Weingarz L, Schwonberg J, Schindewolf M, Hecking C, Wolf Z, Erbe M, Weber A, Lindhoff-Last E, Linnemann B. Prevalence of thrombophilia according to age at the first manifestation of venous thromboembolism: results from the MAISTHRO registry. Br J Haematol. 2013 Dec;163(5):655-65. doi: 10.1111/bjh.12575. Epub 2013 Oct 8. PMID 24219332
- [Result] Kraft C, Hecking C, Schwonberg J, Schindewolf M, Lindhoff-Last E, Linnemann B. Patients with inferior vena cava thrombosis frequently present with lower back pain and bilateral lower-extremity deep vein thrombosis. Vasa. 2013 Jul;42(4):275-83. doi: 10.1024/0301-1526/a000288. PMID 23823859
- [Result] Linnemann B, Meister F, Schwonberg J, Schindewolf M, Zgouras D, Lindhoff-Last E; MAISTHRO registry. Hereditary and acquired thrombophilia in patients with upper extremity deep-vein thrombosis. Results from the MAISTHRO registry. Thromb Haemost. 2008 Sep;100(3):440-6. PMID 18766260
- [Result] Berger M, Moscatelli H, Kulle B, Luxembourg B, Blouin K, Spannagl M, Lindhoff-Last E, Schambeck CM. Association of ADAMDEC1 haplotype with high factor VIII levels in venous thromboembolism. Thromb Haemost. 2008 May;99(5):905-8. doi: 10.1160/TH08-01-0059. PMID 18449420
- [Result] Linnemann B, Schmidt H, Schindewolf M, Erbe M, Zgouras D, Grossmann R, Schambeck C, Lindhoff-Last E. Etiology and VTE risk factor distribution in patients with inferior vena cava thrombosis. Thromb Res. 2008;123(1):72-8. doi: 10.1016/j.thromres.2008.01.004. Epub 2008 Mar 4. PMID 18295303
- [Result] Linnemann B, Zgouras D, Schindewolf M, Schwonberg J, Jarosch-Preusche M, Lindhoff-Last E. Impact of sex and traditional cardiovascular risk factors on the risk of recurrent venous thromboembolism: results from the German MAISTHRO Registry. Blood Coagul Fibrinolysis. 2008 Mar;19(2):159-65. doi: 10.1097/MBC.0b013e3282f54558. PMID 18277138
- [Result] Linnemann B, Schindewolf M, Zgouras D, Erbe M, Jarosch-Preusche M, Lindhoff-Last E. Are patients with thrombophilia and previous venous thromboembolism at higher risk to arterial thrombosis? Thromb Res. 2008;121(6):743-50. doi: 10.1016/j.thromres.2007.07.014. Epub 2007 Sep 4. PMID 17804043